CLINICAL TRIAL: NCT06158087
Title: Prospective, Multicenter, Single-arm Clinical Trial to Evaluate the Safety and Efficacy of pEGASUS Stent System for Assisted Endovascular Treatment of Intracranial Aneurysms
Brief Title: To Evaluate the Safety and Efficacy of Intracranial Stent Assisted Endovascular Treatment of Intracranial Aneurysms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Wallaby Medical Technologies Co.,Inc. (Industry)
Collaborators: Phenox GmbH (Industry); Beijing Wallaby Medical Technologies Co.,Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-1319
Record Dates: First submitted 2023-11-23; First posted 2023-12-06 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2023-11

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): Patients can be included in the study if they meet all of the inclusion and none of the exclusion criteria and have provided written informed consent, intent to use pEGASUS stent system assisted to treat intracranial aneurysm.
  Interventions: Device: pEGASUS Stent System

INTERVENTIONS:
Device: pEGASUS Stent System — Endovascular intervention with p64/p48 MW HPC pEGASUS Stent System was performed in patients diagnosed with intracranial aneurysms

SUMMARY:
The purpose of this study is to assess safety and effectiveness of the pEGASUS stent system.

DETAILED DESCRIPTION:
Title: A prospective, multicenter, single-arm clinical trial to evaluate the safety and efficacy of pEGASUS stent system for assisted endovascular treatment of intracranial aneurysms Device: pEGASUS stent system Design: Prospective, Multicenter, Single Arm Clinical Study. Purpose: To assess safety and effectiveness of the pEGASUS stent system. Study duration: 31 months. Sample Size: 130 patients. Number of sites: ≤10. Follow-up time: 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 80 years, male or female;
* Patients diagnosed as wide-neck intracranial aneurysms by brain CTA/MRA/DSA (neck width≥4mm or bodyor a dome-to-neck ratio<2);
* Parent vessel with a diameter of ≥2.5mm and ≤4.5mm;
* Patients target aneurysm is planned to be embolized using intracranial stent assisted with coiling;
* The mRS Score of the patients was 0-2;
* Patients understand the purpose of the study, accept the follow-up period, and agree to comply with all requirements, agree to participate in the clinical trial and voluntarily sign the informed consent.

Exclusion Criteria:

* Patients who have contraindications to antiplatelet and/or anticoagulant therapy or do not start antiplatelet therapy in time before treatment.
* Patients with anatomical structure is not suitable for endovascular treatment due to severe vascular tortuosity or stenosis shown by angiography.
* Known to be allergic to Nitinol platinum alloy and angiographic agents.
* Conditions that in the opinion of the investigators would prevent patients from completing the study, such as the expected survival period of active tumor less than 1-year, high-risk group of cerebral thrombosis, heart failure and atrial fibrillation.
* Patients combined moyamoya disease, intracranial tumor, intracranial arteriovenous malformation, intracranial arteriovenous fistula and intracranial hematoma.
* The target aneurysm has previously received intravascular embolization or stent implantation treatment;
* Multiple aneurysms or complex aneurysms;
* Patients with acute ruptured aneurysm;
* Serious infection is not controlled and is not suitable for operation;
* Patients who underwent major surgery or interventional therapy (such as brain, cardiac, chest, abdominal or peripheral vascular) within 30 days before surgery;
* Obvious abnormal coagulation function or bleeding tendency;
* Combined with severe renal insufficiency, creatinine greater than or equal to 200umol/L; Patients with severe liver diseases (such as acute and chronic hepatitis, cirrhosis), or ALT more than 3 times the upper normal limit;
* Pregnancy, lactation, or women of childbearing age who plan to be pregnant during the study period;
* Participation in any other clinical trial within 30 days prior to signing informed consent;
* Other conditions considered by the investigator to be inappropriate for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Aneurysm Occlusion of the Treated Target Lesion on 6 Month Angiography | 6 months
  Complete aneurysm occlusion (100% occlusion - Raymond Class 1) of the treated target lesion on 6 month angiography, in the absence of retreatment, or parent artery stenosis (> 50%) at the target location.
Rate of major ipsilateral stroke or neurological death | 12 months
  Any major ipsilateral stroke or neurological death

SECONDARY OUTCOMES:
Technical success rate | Within 24 hours after surgery
  Technical success is defined as the successful placement of pEGASUS stent system.
Rate of successful occlusion | Within 24 hours after surgery, 6 months, 12 months
  Aneurysm successful occlusion is defined as Raymond Grade I/II.
Rate of complete occlusion | Within 24 hours after surgery, 6 months, 12 months
  Aneurysm complete occlusion is defined as Raymond Grade I.
Rate of good clinical prognosis | 3 months, 6 months, 12 months
  Good clinical prognosis means mRS 0~2
Death, stroke, and thrombotic events | to 12 months
  Record the number of death, stroke and thrombotic events throughout the clinical trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No